CLINICAL TRIAL: NCT06364033
Title: Biological and Clinical Efficacy of Recombinant Zoster Vaccine (Shingrix) in Patients With Chronic Lymphocytic Leukemia
Brief Title: Biological and Clinical Efficacy of Shingrix in Patients With CLL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CLL2624
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; CLL-like MBL; Varicella-zoster Virus Reactivation
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: serologic response evaluation — Blood samples collection

SUMMARY:
This is a biological study. Patients who are eligible to receive Shingrix through the Italian National Health System will be invited to participate in the study. According to AIFA indication, the two doses of vaccine will be administered 4-8 weeks apart. Blood samples will be collected prior to the first vaccine dose (i.e. within the time frame of 3 months prior to the first dose) and 1, 6, 12, 24 and 36 months after the second vaccine dose to evaluate the serological response of Shingrix.

DETAILED DESCRIPTION:
This is a multi-centre, prospective study, performed on biological samples only. Patients who are eligible to receive Shingrix through the Italian National Health System will be invited to participate in the study.

According to AIFA indication, the two doses of vaccine will be administered 4-8 weeks apart.

Blood samples will be collected prior to the first vaccine dose (i.e. within the time frame of 3 months prior to the first dose) and 1, 6, 12, 24 and 36 months after the second vaccine dose to evaluate the serological response of Shingrix. All protocol procedures (including clinical assessment and blood draws) will be performed during regular follow-up visits according to clinical practice. No additional invasive/dangerous/painful procedures will be required by the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL or small lymphocytic lymphoma (SLL) or CLL-like MBL according to IWCLL guidelines. Patients must belong to one of the following subgroups:

  * Group A: Patients with MBL or previously untreated early-phase CLL/SLL (Binet stage A or RAI stage 0), with no clear signs of disease progression;
  * Group B: Patients with active or symptomatic disease according to IWCLL guidelines or with advanced Binet or Rai stages receiving both the first and second vaccine doses before treatment initiation;
  * Group C: Patients with CLL/SLL receiving targeted drugs (i.e. ibrutinib/acalabrutinib-based treatment or venetoclax-based treatment) for at least 6 months prior to the administration of the first vaccine dose.
* Age 18 years or older
* Eligible to receive Shingrix according to clinical indication and free of charge through the Italian National Health System
* Life expectancy >6 months
* No active, symptomatic herpes zoster infection or varicella-zoster virus reactivation within 12 months prior to vaccination
* No prior exposure to Shingrix
* Able and willing to provide written informed consent and to comply with the study protocol procedures

Exclusion Criteria:

* Female patients who are currently in pregnancy or are willing to be pregnant
* Any uncontrolled active systemic infection
* Intravenous immunoglobulin (IVIG) administration within 3 months prior to vaccination
* Concomitant use of radiotherapy or chemotherapy
* Hereditary or acquired immunodeficiency syndrome unrelated to CLL
* Chronic use of immunosuppressive medications given for indications that are not CLL-related

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Serologic response evaluation | at 1 month
  Rate of positive serologic response to Shingrix in different subsets of patients as determined by antibody response to varicella-zoster virus (≥4-fold increase in anti-gE titer from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Coscia, Principal Investigator — UOC Ematologia ASST Sette Laghi Varese
Locations (1):
- UOC Ematologia ASST dei Sette Laghi, Varese, Italy